CLINICAL TRIAL: NCT07091981
Title: Effect of Number of Rotary Instruments on Negotiating Second Mesiobuccal Canals to Working Length and on Postoperative Pain: A Randomized Clinical Trial
Brief Title: Effect of Rotary File Number on MB2 Canal Negotiation and Postoperative Pain
Acronym: MB2-PAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Adıgüzel (Other)
Responsible Party: Sponsor-Investigator, Mehmet Adıgüzel, Associate Professor, Mustafa Kemal University
Organization: Mustafa Kemal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HMKU-MB2Pain-RCT2025; 2025/M08-D38 (Other: Hatay Mustafa Kemal Univ EC)
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Pain; Pulp Necrosis
Keywords: VAS Pain Scale; Endodontic Treatment; Rotary Files
MeSH Terms: conditions — Pain, Postoperative; Dental Pulp Necrosis

STUDY DESIGN:
Intervention Model Description: Four parallel arms comparing single-, two-, three-, and four-file rotary systems in maxillary molar canals
Who Masked: Participant
Masking Description: Participants were blinded to the number of rotary instruments used during the root canal procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single-file rotary instrumentation (One Curve) (Experimental): Patients received root canal treatment using a single-file rotary system (OneCurve) in the MB2 canals of maxillary first molars. OneCurve 25/.04 rotary file was used at 300 rpm and 2.5 Ncm torque.
  Interventions: Device: OneCurve Rotary File
- Two-file rotary instrumentation (Perfect Minimally Invasive) (Experimental): Root canal treatment was performed using a two-file system (Perfect Minimally Invasive; Perfect Medical Instruments Co. Ltd, China). A 10/.06 Shaper file was used with brushing motion in the coronal and middle thirds, followed by a 25/.04 Finisher file in the apical third. Files operated at 300 rpm and 2.0-2.5 Ncm torque under continuous irrigation.
  Interventions: Device: Perfect Minimally Invasive Kit
- Three-file rotary instrumentation (VDW Rotate) (Experimental): Root canal instrumentation was performed using a three-file system (VDW Rotate; VDW GmbH, Germany). Instrumentation was performed sequentially using 15/.04, 20/.05, and 25/.04 files for the coronal, middle, and apical thirds, respectively, with brushing-pecking motions in 2-3 mm increments under continuous irrigation. Files were operated at 300 rpm and 1.8 Ncm torque in the MB2 canal of maxillary first molars.
  Interventions: Device: VDW Rotate
- Four-file rotary instrumentation (Perfect Advanced Kit) (Experimental): Root canal instrumentation was performed using a four-file rotary system (Perfect Advanced Kit; Perfect Medical Instruments Co. Ltd, China). Coronal enlargement was initiated with a 10/.07 Opener file at 300 rpm and 2.5 Ncm torque. A 10/.04 file was then used at 250 rpm and 2.0 Ncm torque to reach the apical third. Final shaping was completed with 17/.05 and 25/.04 files at 300 rpm and 2.5 Ncm torque. A crown-down technique was applied using brushing-pecking motions in 2-3 mm increments. After each file, the canal was irrigated thoroughly and file flutes were cleaned to prevent debris accumulation.
  Interventions: Device: Perfect Advanced Kit

INTERVENTIONS:
Device: OneCurve Rotary File — A single-file NiTi system (25/.04) operated at 300 rpm and 2.5 Ncm torque. Applied directly to the MB2 canal without prior hand instrumentation.
  Arms: Single-file rotary instrumentation (One Curve)
Device: Perfect Minimally Invasive Kit — Two-file system using 10/.06 Shaper for coronal/middle thirds and 25/.04 Finisher for apical third. Operated at 300 rpm and 2.0-2.5 Ncm torque.
  Arms: Two-file rotary instrumentation (Perfect Minimally Invasive)
Device: VDW Rotate — Three-file NiTi rotary system (15/.04, 20/.05, 25/.04) used sequentially for coronal, middle, and apical thirds. Applied with brushing-pecking motion in 2-3 mm increments under continuous irrigation. Operated at 300 rpm and 1.8 Ncm torque.
  Arms: Three-file rotary instrumentation (VDW Rotate)
Device: Perfect Advanced Kit — NiTi rotary file system including 10/.07 Opener, 10/.04, 17/.05, and 25/.04 files. Used in crown-down sequence with rpm and torque settings ranging from 250-300 rpm and 2.0-2.5 Ncm. Brushing-pecking motion and continuous irrigation were applied during instrumentation.
  Arms: Four-file rotary instrumentation (Perfect Advanced Kit)

SUMMARY:
This randomized controlled clinical trial aims to evaluate the effect of the number of rotary files on working length negotiation and postoperative pain in the second mesiobuccal (MB2) canals of maxillary first molars. Patients are assigned to one of four groups according to the number of rotary files used: single-, two-, three-, or four-file systems. Postoperative pain is assessed on each of the seven consecutive postoperative days (Days 1-7) using a visual analog scale (VAS), and working length negotiation success is recorded during canal instrumentation.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals aged between 20 and 65 years
* Requiring primary endodontic treatment of maxillary first molars
* Diagnosis of asymptomatic apical periodontitis and pulp necrosis based on clinical and radiographic findings
* Presence of a second mesiobuccal (MB2) canal in the maxillary first molar
* Absence of or only minimal preoperative pain or symptoms
* Periapical lesions smaller than 5 mm in diameter
* Ability to comply with follow-up visits and effectively communicate during the treatment process

Exclusion Criteria:

* Presence of symptomatic apical periodontitis or acute apical abscess
* Retreatment cases (teeth previously treated endodontically)
* Use of medications such as narcotics, antibiotics, sedatives, or antidepressants within one week prior to treatment
* Presence of a sinus tract, periapical abscess, or facial cellulitis
* Pregnancy or breastfeeding
* Inability to understand or follow the study instructions

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-05 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity (VAS Score) | Daily assessment for 7 consecutive days following treatment (Days 1-7)
  Postoperative pain will be assessed using a 100-mm Visual Analog Scale (VAS), where 0 mm represents "no pain" and 100 mm represents "worst possible pain imaginable."

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal University Faculty of Dentistry, Antakya, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) including pain scores (VAS values), demographic data (age, sex), treatment group allocation, and working length negotiation success will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will be available starting from 6 months after study completion (March 2026) and will remain available for 5 years (until March 2031).
Access Criteria: Access will be granted to qualified researchers upon reasonable request. Applicants must submit a proposal outlining the research objectives and intended data use. Data will be shared via secure electronic transfer after approval by the principal investigator. Use is restricted to academic and non-commercial research purposes only.
URL: https://mustafakemal.edu.tr/ipd-sharing-info